CLINICAL TRIAL: NCT02322918
Title: BC Psychosis Program Biobank and Database for Investigating Genetic Polymorphisms of Brain-derived Neurotrophic Factor and Catechol-o-methyl Transferase and Their Associations With Psychosis Disorder
Brief Title: The BC Psychosis Program Biobank and Database for Genetic Polymorphisms and Their Associations With Psychosis Disorder
Acronym: BCPP BIODA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: H14-01136
Record Dates: First submitted 2014-12-12; First posted 2014-12-23 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Psychosis; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — We will be collecting and retaining whole blood samples and saliva samples for genomic testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants admitted to BCPP: Blood or saliva samples will be collected from participants for whole genomic/transcriptomic sequencing
  Interventions: Genetic: Blood samples for whole genomic/transcriptomic sequencing

INTERVENTIONS:
Genetic: Blood samples for whole genomic/transcriptomic sequencing — Participant will receive one blood draw whereby two samples will be extracted. If the participant wishes to participate in the study but is fearful of needles, they may be given the option to provide a saliva sample. A retrospective medical chart review will be performed after participant is discharged from BCPP in order to obtain a full phenotype. Genotyping of BDNF and COMT will be performed. Protein levels of BDNF will be determined. The remaining blood or saliva samples will be stored over the long-term in a biorepository at the BC Mental Health and Addictions Research Institute. A retrospective medical chart review will be completed after the participant is discharged.

SUMMARY:
The purpose of this study is to determine if candidate polymorphisms in brain-derived neurotrophic factor (BDNF) and catechol-o-methyl transferase (COMT) are predictive of psychosis disorder severity, symptomology, and resolution in patients at BCPP. A secondary objective will be to form a biorepository of blood and saliva samples from patients at BCPP so that further genetic, proteonomic and pharmacogenomic studies may be done to gain insight into the genetic basis of differences in psychosis disorder presentation and manifestation, and differences in response to antipsychotic drug treatment.

DETAILED DESCRIPTION:
This is a population-based, genetic-association, candidate polymorphism study. It will involve a prospective and a retrospective component. A blood draw or saliva sample will be performed during the participant's admission to BCPP, which may occur at any point during the participant's length of stay. When a participant has been deemed 'Ready for Discharge' by his/her attending psychiatrist at BCPP, a full phenotype will be obtained via retrospective chart review. Genetic analyses and determination of protein levels will be performed after chart review. Following fulfillment of the primary study objective, the remaining blood and saliva samples will be stored in the biobank over the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Admission to BCPP.
* Has provided written informed consent.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include all patients who have been admitted to the British Columbia Psychosis Program (BCPP). BCPP provides intensive inpatient care for individuals who have psychosis-related treatment challenges, including pharmacologic, biophysical, and psychosocial services. Admission criteria to BCPP include the following: 1) Must be 18 years or older; 2) Diagnosis of schizophrenia, schizoaffective disorder, mood disorder with psychosis; 3) History of no response or inadequate response of positive symptoms to at least 2 adequate trials of antipsychotics (one of which is a second generation agent) by health authority tertiary clinical teams; 4) Incomplete recovery of social, vocational, and occupational functioning and 5) If present, substance use disorder, pervasive developmental disorder, developmental disability, personality disorder, aggression, or head injury are not the primary focuses of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Creation of biorepository of blood samples for future genetic, proteonomic and pharmacogenomic studies. | One visit during participant's stay at BCPP, an expected average of 6 months
  A biobank of stored samples will be used to determine the genetic variability in psychosis disorder.

SECONDARY OUTCOMES:
Identification of single-nucleotide polymorphisms (SNPs) in the BDNF and COMT genes | One visit during participant's stay at BCPP, an expected average of 6 months
  We will determine if specific genetic variants in BDNF and COMT genes are associated with psychosis disorder severity, symptomology and resolution.
Medical Chart Review | One visit during participant's stay at BCPP, an expected average of 6 months
  A medical chart review will be done on hard-copy medical charts at BCPP.

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair M Barr, Ph.D., Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Hospital - BC Psychosis Program, Vancouver, British Columbia, Canada